CLINICAL TRIAL: NCT01896102
Title: A Phase 2/3 Study of the Efficacy and Safety of Hematopoietic Stem Cells Transduced With Lenti-D Lentiviral Vector for the Treatment of Cerebral Adrenoleukodystrophy (CALD)
Brief Title: A Study of the Efficacy and Safety of Hematopoietic Stem Cells Transduced With Lenti-D Lentiviral Vector for the Treatment of Cerebral Adrenoleukodystrophy (CALD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALD-102; 2011-001953-10 (EudraCT Number)
Record Dates: First submitted 2013-03-22; First posted 2013-07-11 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Adrenoleukodystrophy (CALD)
Keywords: Adrenoleukodystrophy; X-linked adrenoleukodystrophy; Gene therapy; Hematopoietic stem cell
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenti-D Drug Product (Experimental): Participants received a single intravenous (IV) infusion of Lenti-D Drug Product at a dose of greater than or equal to (>=) 5.0 × 10^6 CD34+ cells/kilogram (kg) (autologous CD34+ cell-enriched population that contained cells transduced with lentiviral vector encoding ABCD1 cDNA for human adrenoleukodystrophy protein, suspended in a cryopreservative solution) on Day 0.
  Interventions: Genetic: Lenti-D Drug Product (eli-cel)

INTERVENTIONS:
Genetic: Lenti-D Drug Product (eli-cel) — Participants received a single IV infusion of Lenti-D Drug Product.
  Other Names: elivaldogene autotemcel; eli-cel

SUMMARY:
This trial assessed the efficacy and safety of autologous cluster of differentiation 34 (CD34+) hematopoietic stem cells, transduced ex-vivo with Lenti-D lentiviral vector (also called elivaldogene autotemcel or eli-cel), for the treatment of cerebral adrenoleukodystrophy (CALD). A participant's blood stem cells were collected and modified (transduced) using the Lenti-D lentiviral vector encoding human adrenoleukodystrophy protein. After modification (transduction) with the Lenti-D lentiviral vector, the cells were transplanted back into the participant following myeloablative conditioning. Participants in this study will be continuously followed in study LTF-304.

DETAILED DESCRIPTION:
For study ALD-102 the Transplant Population (TP), Neutrophil Engraftment Population (NEP), and Intent-to-Treat Population (ITT) were identical.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent was obtained from a competent custodial parent or guardian with legal capacity to execute a local institutional review board (IRB)/Independent Ethics Committee (IEC) approved consent (informed assent will be sought from capable participants, in accordance with the directive of the IRB/IEC and with local requirements).
2. Males aged 17 years and younger, at the time of parental/guardian consent and, where appropriate, participant assent.
3. Active cerebral adrenoleukodystrophy (ALD) as defined by:

   1. Elevated very long chain fatty acids (VLCFA) values, and
   2. Active CNS disease established by central radiographic review of brain magnetic resonance imaging (MRI) demonstrating:
   3. Loes score between 0.5 and 9 (inclusive) on the 34-point scale, and
   4. Gadolinium enhancement on MRI of demyelinating lesions.
4. NFS less than or equal to (<or=) 1.

Exclusion Criteria:

1. Receipt of an allogeneic transplant or gene therapy.
2. Availability of a willing 10/10 HLA-matched sibling donor (excluding female heterozygotes).
3. Use of statins, Lorenzo's Oil, or dietary regimens used to lower very long chain fatty acids (VLCFA) levels. Note: participants must discontinue use of these medications at time of consent.
4. Receipt of an investigational study drug or procedure within 3 months before Screening that might confound study outcomes. Use of investigational study drugs is prohibited throughout the course of the study.
5. Any conditions that make it impossible to perform MRI studies (including allergies to anesthetics or contrast agents).
6. Hematological compromise as evidenced by:

   * Peripheral blood absolute neutrophil count (ANC) count < 1500 cells/ cubic milli meter (mm3),
   * Platelet count < 100,000 cells/mm3, or
   * Hemoglobin < 10 gram per deciliter (g/dL).
   * Uncorrected bleeding disorder.
7. Hepatic compromise as evidenced by:

   * Aspartate transaminase (AST) value > 2.5×upper limit of normal (ULN)
   * Alanine transaminase (ALT) value > 2.5×ULN
   * Total bilirubin value > 3.0 milligram per deciliter (mg/dL), except if there is a diagnosis of Gilbert's Syndrome and the participant is otherwise stable
8. Renal compromise as evidenced by abnormal renal function (actual or calculated creatinine clearance < 50 milliliter per minute [mL/min])
9. Cardiac compromise as evidenced by left ventricular ejection fraction <40 percent (%)
10. Immediate family member with a known or suspected Familial Cancer Syndrome (including but not limited to hereditary breast and ovarian cancer syndrome, hereditary non-polyposis colorectal cancer syndrome, and familial adenomatous polyposis).
11. Clinically significant active bacterial, viral, fungal, parasitic, or prion-associated infection
12. Positive for human immunodeficiency virus type 1 or 2 (HIV-1, HIV-2); hepatitis B; hepatitis C; human T lymphotrophic virus 1 (HTLV-1). (Note that participants who have been vaccinated against hepatitis B [hepatitis B surface antibody-positive] who are negative for other markers of prior hepatitis B infection [eg, negative for hepatitis B core antibody (Ab)] are eligible. Participants with past exposure to hepatitis B virus (HBV [HBcAb positive and/or HBeAb positive]) are also eligible for the study provided they have a negative test for HBV DNA. Also note that participants who are positive for anti-hepatitis C antibody are eligible as long as they have a negative hepatitis C viral load.
13. Any clinically significant cardiovascular or pulmonary disease, or other disease or condition that would be contraindicated for any of the other study procedures.
14. Absence of adequate contraception for fertile participants. Male participants and their female partners are required to use two different effective methods of contraception from Screening through at least 6 months after drug product infusion. If subjects are truly sexually abstinent (where true sexual abstinence is defined as being in line with the preferred and usual lifestyle of the subject), no second method is required.
15. Any contraindications to the use of granulocyte colony stimulating (G-CSF) during the mobilization of HSCs, and any contraindications to the use of busulfan or cyclophosphamide, including known hypersensitivity to the active substances or to any of the excipients in their formulations.

Max Age: 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2013-08-21 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Sieker, MD., Study Director — bluebird bio, Inc.; David Williams, MD, Principal Investigator — Boston Children's Hospital; Christine Duncan, MD, Principal Investigator — Boston Children's Hospital; Florian Eichler, MD, Principal Investigator — Massachusetts General Hospital; Satiro de Oliveira, MD, Principal Investigator — University of California, Los Angeles; Paul Orchard, MD, Principal Investigator — University of Minnesota; Adrian Thrasher, MD, PhD, Principal Investigator — Great Ormond Street Hospital for Chidren NHS Foundation Trust; Patrick Aubourg, MD, PhD, Principal Investigator — Hôpital Bicêtre; Jorn-Sven Kuhl, MD, Principal Investigator — University of Leipzig; Nicholas Smith, MD, Principal Investigator — Women and Children's Hospital; Hernan Amartino, MD, Principal Investigator — Medeos SRL
Locations (8):
- United States (3):
  - Mattel Children's Hospital UCLA/Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Boston Children's Hospital/Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
- Medeos SRL, Buenos Aires, Argentina
- Women and Children's Hospital, North Adelaide, South Australia, Australia
- Hôpital Bicêtre, Le Kremlin-Bicêtre, France
- University of Leipzig, Leipzig, Germany
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Bluebird bio is committed to transparency and appropriately de-identified patient-level datasets and supporting documents may be shared following attainment of applicable marketing approvals associated with this study and consistent with criteria established by bluebird bio and/or industry best practices to maintain the privacy of study participants. Note that given the rarity of the disease and the identifiable nature of the participants in this study, it is anticipated that the sharing of data from this study may be limited. For enquiries, please contact us at datasharing@bluebirdbio.com.

REFERENCES:
- [Derived] Eichler F, Duncan CN, Musolino PL, Lund TC, Gupta AO, De Oliveira S, Thrasher AJ, Aubourg P, Kuhl JS, Loes DJ, Amartino H, Smith N, Folloni Fernandes J, Sevin C, Sankar R, Hussain SA, Gissen P, Dalle JH, Platzbecker U, Downey GF, McNeil E, Demopoulos L, Dietz AC, Thakar HL, Orchard PJ, Williams DA. Lentiviral Gene Therapy for Cerebral Adrenoleukodystrophy. N Engl J Med. 2024 Oct 10;391(14):1302-1312. doi: 10.1056/NEJMoa2400442. PMID 39383459
- [Derived] Duncan CN, Bledsoe JR, Grzywacz B, Beckman A, Bonner M, Eichler FS, Kuhl JS, Harris MH, Slauson S, Colvin RA, Prasad VK, Downey GF, Pierciey FJ, Kinney MA, Foos M, Lodaya A, Floro N, Parsons G, Dietz AC, Gupta AO, Orchard PJ, Thakar HL, Williams DA. Hematologic Cancer after Gene Therapy for Cerebral Adrenoleukodystrophy. N Engl J Med. 2024 Oct 10;391(14):1287-1301. doi: 10.1056/NEJMoa2405541. PMID 39383458
- [Derived] Eichler F, Duncan C, Musolino PL, Orchard PJ, De Oliveira S, Thrasher AJ, Armant M, Dansereau C, Lund TC, Miller WP, Raymond GV, Sankar R, Shah AJ, Sevin C, Gaspar HB, Gissen P, Amartino H, Bratkovic D, Smith NJC, Paker AM, Shamir E, O'Meara T, Davidson D, Aubourg P, Williams DA. Hematopoietic Stem-Cell Gene Therapy for Cerebral Adrenoleukodystrophy. N Engl J Med. 2017 Oct 26;377(17):1630-1638. doi: 10.1056/NEJMoa1700554. Epub 2017 Oct 4. PMID 28976817
- See also: ALD-102 is parent study for LTF-304 study — https://clinicaltrials.gov/show/NCT02698579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 centers from 21 August 2013 (first participants first visit) to 26 March 2021 (last participants last visit).
Pre-assignment Details: A total of 32 Participants were enrolled and treated in this study. All male participants with Cerebral Adrenoleukodystrophy (CALD) were treated with Lenti-D Drug Product also referred to as eli-cel (elivaldogene autotemcel) in this study. For study ALD-102 the Transplant Population (TP), Neutrophil Engraftment Population (NEP), and Intent-to-Treat Population (ITT) are identical.
Groups:
- Lenti-D Drug Product: Participants received a single intravenous (IV) infusion of Lenti-D Drug Product at a dose of greater than or equal to (>=) 5.0 × 10^6 CD34+ cells/kilogram (kg) (autologous CD34+ cell-enriched population that contains cells transduced with lentiviral vector encoding ABCD1 cDNA for human adrenoleukodystrophy protein, suspended in a cryopreservative solution) on Day 0. Neutrophil Engraftment Population (NEP) is identical to the Transplant Population (TP).
Period: Overall Study
Arm/Group | Lenti-D Drug Product
Started | 32
Completed | 29
Not Completed | 3
Not completed — Death | 1
Not completed — Participant to receive allogenic transplant | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat Population (ITT) consisted of participants who initiated any study procedures, beginning with mobilization by granulocyte colony-stimulating factor (G-CSF).
Groups:
- Lenti-D Drug Product: Participants received a single intravenous (IV) infusion of Lenti-D Drug Product at a dose of greater than or equal to (>=) 5.0 × 10^6 CD34+ cells/kilogram (kg) (autologous CD34+ cell-enriched population that contains cells transduced with lentiviral vector encoding ABCD1 cDNA for human adrenoleukodystrophy protein, suspended in a cryopreservative solution) on Day 0.
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 5
  Unknown or Not Reported | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Alive and Have None of the 6 Major Functional Disabilities (MFDs) at Month 24 and Without Allo-HSCT or Rescue Cell Administration
Description: The 6 MFDs consisted of loss of communication, cortical blindness, tube feeding, total incontinence, wheelchair dependence, complete loss of voluntary movement. Month 24 MFD-Free survival criteria was defined as: alive at 24 months post-infusion; had not developed any of the MFDs by 24 months post-infusion; had not received rescue cell administration or allo-HSCT by 24 months post-infusion; and had not withdrawn from the study or had not been lost to follow-up by 24 months post-infusion. Percentage of participants who were alive and have none of the 6 major functional disabilities (MFDs) at Month 24 were reported.
Time Frame: At Month 24
Population: Transplant Population (TP) consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants were defined as those who had been followed for 24 months (i.e. Rel DLC >= 730) or have had completed Month 24, or discontinued from the study but would have been followed for 24 months if still on the study (i.e. Rel Day of data cut >= 730).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants | 90.6 [75.0 to 98.0]

2. Primary Outcome: Proportion of Participants Who Had Experienced Either Acute ([>or=] Grade II) or Chronic Graft Versus Host Disease (GVHD) by Month 24
Description: Acute GVHD graded on the Acute GVHD Grading Scale (I-IV): Grade I is characterized as mild disease, Grade II as moderate, Grade III as severe (involvement of any organ system), and Grade IV as life-threatening; chronic GVHD was determined by the Investigator. Percentage of participants who experienced with either acute (>= Grade II) or chronic GVHD at Month 24 were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. To be evaluable participants must have either experienced the event by Month 24 (Rel Day 730) or have been followed for at least 12 months (Rel Day of DLC >= 365) without GVHD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants | 0.0 [0.0 to 10.9]

3. Secondary Outcome: Percentage of Participants Who Demonstrated Resolution of Gadolinium Positivity on Magnetic Resonance Imaging (MRI) at Month 24
Description: Percentage of participants who demonstrated resolution of gadolinium positivity (i.e., GdE-) on MRI at Month 24 were reported.
Time Frame: At Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Evaluable participants are defined as participants who completed the Month 24 assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 30
Percentage of participants | 86.7 [69.3 to 96.2]

4. Secondary Outcome: Time to Sustained Resolution of Gadolinium Positivity on MRI
Description: Sustained resolution of gadolinium positivity was defined as having at least two consecutive GdE- results by MRI without a subsequent evaluation indicating GdE+.
Time Frame: Up to Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Here, "Overall Number of participants Analyzed" signifies those participants who were evaluable for this outcome measure. Evaluable participants are defined as participants who have completed the Month 24 assessment of GdE status.
Measure: Median (Full Range); unit: Days
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 24
Days | 77 [25 to 551]

5. Secondary Outcome: Number of Participants With Change in Total Neurologic Function Score (NFS) From Baseline up to Month 24
Description: NFS was a 25-point score used to evaluate the severity of gross neurologic dysfunction in CALD by scoring 15 symptoms (functional domains) across 6 categories. Listed here are the 15 symptoms followed by their maximal score out of 25 points: a) Hearing / auditory processing problems-1, b) Aphasia/apraxia-1, c) Loss of communication-3, d) Vision impairment/field cut-1, e) Cortical blindness-2, f) Swallowing/other CNS dysfunctions-2, g) Tube feeding-2, h) Running difficulties/hyperreflexia-1, i) Walking difficulties/spasticity/spastic gait (no assistance)-1, j) Spastic gait (needs assistance)-2, k) Wheelchair dependence-2, l) Complete loss of voluntary movement-3, m) Episodes of incontinence -1, n) Total incontinence-2, o) Nonfebrile seizures-1. A score of "0" denoted absence of clinical signs of cerebral disease. Maximal signs within a domain score the total of all grades within that domain. Number of participants with change in total NFS from baseline up to Month 24 were reported.
Time Frame: Baseline up to Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Evaluable participants are defined as participants who have non-missing Baseline and have completed the Month 24 NFS assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 30
Participants | 4

6. Secondary Outcome: Major Functional Disability (MFD)-Free Survival Rate
Description: MFD-free survival rate was defined as percentage of participants from drug product infusion to either second transplant, MFD, or death due to any cause, whichever occurs first. MFD-free survival rate was analyzed using Kaplan-Meier Analysis. Kaplan-Meier estimated MFD-free survival rate at 24 months after Lenti-D drug infusion was reported.
Time Frame: At 24 months after Lenti-D drug infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants | 90.6 [73.7 to 96.9]

7. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate was defined as percentage of participants alive from date of Lenti-D drug product infusion (Day 0) to date of death of all causes. Overall survival rate was censored at the date of last visit if the participant were alive. Participants who are alive were censored at the date of last contact. Overall survival rate was analyzed using Kaplan-Meier Analysis. Kaplan-Meier estimated overall survival rate at 24 months after Lenti-D drug infusion was reported.
Time Frame: At 24 months after Lenti-D drug infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants | 96.7 [78.6 to 99.5]

8. Secondary Outcome: Proportion of Participants With Neutrophil Engraftment by 42 Days Post-drug Product Infusion
Description: Neutrophil engraftment (NE) was defined as achieving 3 consecutive absolute neutrophil count (ANC) laboratory values of >= 0.5×10^9 cells/Liter (L) (after initial post-infusion nadir) obtained on different days by 42 days post-infusion of Lenti-D Drug Product (Relative Day 43). Percentage of participants with neutrophil engraftment by 42 Days post-drug product infusion were reported.
Time Frame: By 42 days post-drug infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants for NE if they achieved neutrophil engraftment by Rel Day 43, or had discontinued or were lost to follow-up before Rel Day 43 without achieving NE, or had been followed to at least Rel Day 43 but had not achieved NE. Participants who discontinued or were lost to follow-up before Rel Day 43 without achieving NE were considered failures for NE.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants | 100.0 [89.1 to 100]

9. Secondary Outcome: Time to Neutrophil Engraftment Post-drug Product Infusion
Description: Neutrophil Engraftment was defined as achieving 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion nadir) obtained on different days by 42 days post-infusion of Lenti-D Drug Product (Relative Day 43). Time to neutrophil engraftment post-drug product infusion was reported.
Time Frame: By 42 days post-drug infusion
Population: TP consisted of Participants who received Lenti-D Drug Product infusion. Participants were evaluable for NE if: 1) They achieved Neutrophil Engraftment by Rel Day 43 2)Had discontinued or were lost to follow-up before Rel Day 43 without achieving NE 3) Had been followed to at least Rel Day 43 but had not achieved NE. Participants who discontinued or were lost to follow-up before Rel Day 43 without achieving NE were considered failures for NE.
Measure: Median (Full Range); unit: Days
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Days | 13.0 [11 to 41]

10. Secondary Outcome: Proportion of Participants With Platelet Engraftment by Month 24
Description: Platelet Engraftment was defined as achieving 3 consecutive unsupported platelet counts of >=20 × 10^9 cells/L (after initial post-infusion nadir) obtained on different days while no platelet transfusions were administered for 7 days immediately preceding and during the evaluation period. The first day of 3 consecutive platelet counts >=20 × 10^9 cells/L was the day of PE. Percentage of participants with Platelet Engraftment by Month 24 (Rel Day 730) were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Participants were evaluable for platelet engraftment if they achieved Platelet Engraftment by 24 months (Rel Day 730), or had been followed for at least 24 months without any events.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants | 100 [89.1 to 100.0]

11. Secondary Outcome: Time to Platelet Engraftment Post-drug Product Infusion
Description: Platelet Engraftment was defined as achieving 3 consecutive unsupported platelet counts of > or =20 × 10^9 cells/L (after initial post-infusion nadir) obtained on different days while no platelet transfusions were administered for 7 days immediately preceding and during the evaluation period. The first day of 3 consecutive platelet counts >=20 × 10^9 cells/L was the day of PE. Time to Platelet Engraftment post-drug product infusion up to Month 24 was reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Participants were evaluable for Platelet Engraftment if they had achieved platelet engraftment by 24 months (Rel Day 730), or had been followed for at least 24 months without any events.
Measure: Median (Full Range); unit: Days
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Days | 32 [16 to 60]

12. Secondary Outcome: Proportion of Participants With Engraftment Failure By Month 24
Description: Participants were considered to have primary engraftment failure if they did not achieve NE by Relative Day 43. A participant was considered to have secondary engraftment failure if they achieved and then subsequently lost NE by the Month 24, i.e., if they met both the conditions; Achieved NE by Relative Day 43 as defined above and had sustained decline in ANC to < 0.5×10^9 cells/L for 3 consecutive measurements on different days after Relative Day 43, without alternate etiology. First day of the 3 consecutive ANC decline to < 0.5×10^9 cells/L was considered the day of secondary engraftment failure. Percentage of participants with both primary and secondary engraftment failure at Month 24 were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Here, "Overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. Evaluable participants for secondary Neutrophil Engraftment failure included participants who had achieved neutrophil engraftment, and 1) have secondary engraftment failure by Rel Day 730, or 2) had been followed for at least 24 months without any events.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 29
Percentage of participants | 0.0 [0.0 to 11.9]

13. Secondary Outcome: Proportion of Participants Who Underwent a Subsequent Allo-Hematopoietic Stem Cell (HSC) Infusion by Month 24
Description: Percentage of Participants who have undergone a subsequent allo-HSC infusion at Month 24 were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Evaluable participants were defined as those who decided to receive subsequent allo-HSCT thus discontinued from the study, or participants who have been followed for at least 24 months (Rel Day of last contact >= 730 or completed Month 24 visit) if no events.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 31
Percentage of participants | 6.5 [0.8 to 21.4]

14. Secondary Outcome: Percentage of Participants With Transplant-related Mortality Through 100 and 365 Days Post-drug Product Infusion
Description: Transplant-related mortality was determined by the Investigator in participants who had died from transplant-related causes by 100 days post-drug product infusion (Rel Day 101) or 365 days post-drug product infusion (Rel Day 366) respectively or had been followed to at least Rel Day 101 or 366 respectively if no events yet. Percentage of participants with transplant-related mortality through 100 and 365 days post-drug product infusion were reported.
Time Frame: From time of drug product infusion through 100 and 365 days post-drug product infusion
Population: TP consisted of participants who received Lenti-D Drug Product infusion. Evaluable participants included participants who had died from transplant-related causes by Rel Day 101 or 366 respectively or have been followed to at least Rel Day 101 or 366 respectively if no events yet.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants
  Transplant-related mortality within 100 days | 0.0 [0.0 to 10.9]
  Transplant-related mortality within 365 days | 0.0 [0.0 to 10.9]

15. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious AEs, Grade >=3 AE, Related AEs, Related SAEs and Related Grade >=3 AEs
Description: Adverse event was defined as any untoward medical occurrence associated with the use of a drug product in participants, whether or not considered drug related. SAE was any AE, occurring at any dose and regardless of causality, that resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or was considered an important medical event that may jeopardize the participant and may require medical or surgical intervention to prevent an outcome listed previously. Percentage of participants with all AEs, all SAEs, all drug-product related AEs and SAEs Grade >=3 (severe or medically significant but not immediately life threatening AE) and related Grade >=3 AEs were reported.
Time Frame: From date of informed consent up to Month 24
Population: ITT population consisted of participants who initiated any study procedures, beginning with mobilization by G-CSF
Measure: Number; unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants
  Percentage of participants with at least 1 AE | 100.0
  Percentage of participants with at least 1 SAE | 65.6
  Percentage of participants with at least 1 AE related to Lenti-D Drug | 9.4
  Percentage of participants with at least 1 SAE related to Lenti-D Drug | 3.1
  Percentage of participants with at least 1 Grade >=3 AE | 93.8
  Percentage of participants with at least 1 Grade>=3 AE related to Lenti-D Drug | 3.1

16. Secondary Outcome: Percentage of Participants With Potentially Clinical Significant Changes in Laboratory Parameters by Month 24
Description: Laboratory parameters included hematology (Leukocytes [with a threshold (TS) range <4.0 x 10^9/L, >=18 x 10^9/L], Neutrophils [<1.0 x 10^9/L], Erythrocytes [<=3.0 x 10^12/L], Platelets [<=75 x 10^9/L]); clinical chemistry (Sodium [<=126 millimoles per liter (mmol/L), >=156 mmol/L], Potassium [<=3 mmol/L, >=6 mmol/L], Glucose [<=3.0 mmol/L], Urea Nitrogen [>=10.7 mmol/L], Creatinine [>=150 umol/L]) and liver function tests (LFT) (Alanine Aminotransferase [ALA]. Aspartate Aminotransferase [ASA], Alkaline Phosphatase [AP] with TS range of >=3 x upper limit of normal (ULN), Bilirubin [>=34.2 micromoles per liter (umol/L)]). Clinical significance was decided by investigator.
Time Frame: From time of drug product infusion up to Month 24
Population: ITT population consisted of participants who initiated any study procedures, beginning with mobilization by G-CSF.
Measure: Number; unit: Percentage of participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Percentage of participants
  Hematology: Leukocytes (<4.0 x 10^9/L) | 100.0
  Hematology: Leukocytes (>=18 x 10^9/L) | 0.0
  Hematology: Neutrophils (<1.0 x 10^9/L) | 78.1
  Hematology: Erythrocytes (<=3.0 x 10^12/L) | 43.8
  Hematology: Platelets (<=75 x 10^9/L) | 96.9
  Chemistry: Sodium (<=126 mmol/L) | 0.0
  Chemistry: Sodium (>=156 mmol/L) | 0.0
  Chemistry: Potassium (<=3 mmol/L) | 21.9
  Chemistry: Potassium (>=6 mmol/L) | 0.0
  Chemistry: Glucose (<=3.0 mmol/L) | 0.0
  Chemistry: Urea Nitrogen (>=10.7 mmol/L) | 0.0
  Chemistry: Creatinine (>=150 umol/L) | 0.0
  LFT: ALA (>=3 x ULN) | 3.1
  LFT: ASA (>=3 x ULN) | 3.1
  LFT: AP (>=3 x ULN) | 0.0
  LFT: Bilirubin (>=34.2 umol/L) | 0.0

17. Secondary Outcome: Number of Emergency Room Visits (Post-Neutrophil Engraftment) By Month 24
Description: Number of emergency room visits (post-neutrophil engraftment) up to Month 24 were reported.
Time Frame: From Post-Neutrophil Engraftment up to Month 24
Population: The successful Neutrophil Engraftment Population (NEP) consisted of participants who achieved NE defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion) obtained on different days of post-infusion of Lenti-D Drug Product.
Measure: Number; unit: Emergency room visits
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Emergency room visits | 13

18. Secondary Outcome: Number of In-patient Hospitalizations (Post-Neutrophil Engraftment) By Month 24
Description: Number of In-patient hospitalizations (post-neutrophil engraftment) by Month 24 were reported.
Time Frame: From post-neutrophil engraftment up to Month 24
Population: The successful NEP consisted of participants who achieved NE defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion) obtained on different days of post-infusion of Lenti-D Drug Product.
Measure: Number; unit: Hospitalizations
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Hospitalizations | 14

19. Secondary Outcome: Duration of In-patient Hospitalizations (Post-Neutrophil Engraftment) up to Month 24
Description: Duration of in-patient hospitalizations was calculated as: Duration = (Date of hospital discharge) - (Date of hospital admission before NE) + 1. Duration of In-patient hospitalizations (post-neutrophil engraftment) up to Month 24 was reported.
Time Frame: From post-neutrophil engraftment up to Month 24
Population: The successful NEP consisted of participants who achieved NE defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion) obtained on different days of post-infusion of Lenti-D Drug Product. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 14
Days | 3.0 [2 to 33]

20. Secondary Outcome: Number of Intensive Care Units (ICU) Stays (Post-neutrophil Engraftment) By Month 24
Description: Number of ICU Stays (Post-neutrophil Engraftment) By Month 24 were reported.
Time Frame: From post-neutrophil engraftment up to Month 24
Population: The successful NEP consisted of participants who achieved NE defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion) obtained on different days by of post-infusion of Lenti-D Drug Product.
Measure: Number; unit: ICU Stays
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
ICU Stays | 1

21. Secondary Outcome: Duration of ICU Stays (Post-neutrophil Engraftment) By Month 24
Description: Duration of ICU Stays was calculated as: Duration = (Date of hospital discharge) - (Date of hospital admission before NE) + 1. Duration of ICU Stays (Post-neutrophil Engraftment) by Month 24 was reported.
Time Frame: From post-neutrophil engraftment up to Month 24
Population: The successful NEP consisted of participants who achieved NE defined as having 3 consecutive ANC laboratory values of >= 0.5×10^9 cells/L (after initial post-infusion) obtained on different days of post-infusion of Lenti-D Drug Product. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 1
Days | 12.0 [12 to 12]

22. Secondary Outcome: Number of Participants With Vector-Derived Replication Competent Lentivirus (RCL) Detected by Month 24
Description: Number of Participants with Vector-derived RCL detected at Month 24 were reported. Screening participants blood samples for RCL at month 24 following Lenti-D Drug infusion was performed, with the more rigorous co-culture assays used to distinguish any false positives as applicable.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Participants | 0

23. Secondary Outcome: Number of Participants With Insertional Oncogenesis By Month 24
Description: Insertional oncogenesis including myelodysplasia, leukemia, lymphoma. Number of participants with insertional oncogenesis at Month 24 were reported.
Time Frame: By Month 24
Population: TP consisted of participants who received Lenti-D Drug Product infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenti-D Drug Product
Number analyzed (Participants) | 32
Participants | 0

ADVERSE EVENTS:
Time Frame: From date of informed consent up to Month 24
Arm/Group | Lenti-D Drug Product
All-Cause Mortality (participants affected / at risk) | 1/32
Serious Adverse Events (participants affected / at risk) | 21/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenti-D Drug Product (N=32)
Pyrexia (General disorders) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Vascular device infection (Infections and infestations) | 3 (3)
Cystitis viral (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Neurological decompensation (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenti-D Drug Product (N=32)
Thrombocytopenia (Blood and lymphatic system disorders) | 31 (31)
Anaemia (Blood and lymphatic system disorders) | 31 (31)
Neutropenia (Blood and lymphatic system disorders) | 30 (30)
Febrile neutropenia (Blood and lymphatic system disorders) | 20 (20)
Leukopenia (Blood and lymphatic system disorders) | 11 (11)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6)
Bradycardia (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 30 (30)
Vomiting (Gastrointestinal disorders) | 28 (28)
Stomatitis (Gastrointestinal disorders) | 27 (27)
Abdominal pain (Gastrointestinal disorders) | 17 (17)
Diarrhoea (Gastrointestinal disorders) | 14 (14)
Constipation (Gastrointestinal disorders) | 9 (9)
Oral pain (Gastrointestinal disorders) | 3 (3)
Proctitis (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 2 (2)
Pyrexia (General disorders) | 11 (11)
Catheter site pain (General disorders) | 8 (8)
Catheter site hemorrhage (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Vascular device infection (Infections and infestations) | 3 (3)
Enterobiasis (Infections and infestations) | 2 (2)
Oral candiasis (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 7 (7)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Blood creatinine increased (Investigations) | 2 (2)
C-reactive protein increased (Investigations) | 2 (2)
International normalised ratio increased (Investigations) | 2 (2)
Protein total decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 22 (22)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (20)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (9)
Hyphophosphataemia (Metabolism and nutrition disorders) | 5 (5)
Fluid Retention (Metabolism and nutrition disorders) | 4 (4)
Headache (Nervous system disorders) | 13 (13)
Lethargy (Nervous system disorders) | 2 (2)
Sensory loss (Nervous system disorders) | 2 (2)
Visual field defect (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Irritability (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 23 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4)
Rash Maculo papular (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (4)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dystonia (Nervous system disorders) | 2 (2)
Speech disorder (Nervous system disorders) | 2 (2)
Enuresis (Psychiatric disorders) | 3 (3)
Agitation (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Encopresis (Psychiatric disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT01896102/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT01896102/SAP_001.pdf